CLINICAL TRIAL: NCT05596084
Title: Clinical, Radiological and Histological Comparison of the Use of Bovine Bone Graft and Titanium-Platelet Rich Fibrin in Maxillary Sinus Augmentation: Split-Mouth Randomized Controlled Trials
Brief Title: Comparison of the Use of Bovine Bone Graft and Titanium-Platelet Rich Fibrin in Maxillary Sinus Augmentation
Acronym: T-PRF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Principal Investigator, Berceste Guler, Assoc. Prof., Kutahya Health Sciences University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2022-03/05
Record Dates: First submitted 2022-10-23; First posted 2022-10-27 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Sinus Disease; Maxillary Sinus Disease
Keywords: maxillary sinus augmentation; xenograft; platelet-rich fibrin prepared with titanium
MeSH Terms: conditions — Paranasal Sinus Diseases | interventions — Titanium

STUDY DESIGN:
Intervention Model Description: The maxillary sinus augmentation procedure has been a common treatment method since the 1980s. In patients who have insufficient bone height in the maxillary posterior edentulous region and who want implant placement, materials that provide bone formation are placed in the sinus cavity. When the bone height is 4 mm or less, it is necessary to provide bone formation with maxillary sinus augmentation surgery 6 months before implant placement. The aim of this study is to determine the primary stability of the implant by placing a titanium-rich fibrin on one side and a bovine bone graft on the other side with a sinus lift applied 6 months before the implant in bilateral maxillary posterior region with insufficient bone height with tooth deficiency. is the evaluation of the effect on the obtained bone histology, volume, height and density.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bio-oss bovine bone graft with maxillary sinus augmentation and implant placement (Experimental): A 2 cc Bio-oss bovine bone graft will be used for maxillary sinus augmentation before placing an implant on one side of the bilateral atrophic maxillary posterior regions. Then, 6 months after the surgery, the implant will be placed in accordance with the standard protocol
  Interventions: Procedure: Maxillary sinus augmentation with bovine bone graft
- Titanium-Platelet Rich Fibrin with maxillary sinus augmentation and implant placement (Experimental): A Titanium-Platelet Rich Fibrin will be used for maxillary sinus augmentation before placing an implant on other side of the bilateral atrophic maxillary posterior regions. Titanium platelet-rich fibrin was prepared by centrifugation at 2700 rpm for 14 minutes in accordance with standard protocols. Then, 6 months after the surgery, the implant will be placed in accordance with the standard protocol
  Interventions: Procedure: maxillary sinus augmentation and implant placement

INTERVENTIONS:
Procedure: maxillary sinus augmentation and implant placement — For maxillary sinus augmentation, the area will be prepared by lifting a full-thickness flap. The sinus membrane will be carefully elevated by opening a window through the lateral wall of the sinus on both sides.platelet-rich fibrin prepared with titanium on the other side will be placed in the space prepared in the sinus region by random selection. For Platelet-rich fibrin prepared with titanium (T-PRF), the blood taken from the patient to a 20 cc injektor was put into titanium tubes and prepared by centrifugation at 2700 rpm for 14 minutes according to the standard protocol. Then, 6 months after the surgery, histological sample will be taken with a trephine bur in both groups and the implant will be placed in accordance with the standard protocol. The stability value (ISQ) of the placed implant will be measured with the Ostell device at the time the implant is placed and 3 months after it is placed.
  Other Names: Platelet-rich fibrin prepared with titanium
  Arms: Titanium-Platelet Rich Fibrin with maxillary sinus augmentation and implant placement
Procedure: Maxillary sinus augmentation with bovine bone graft — For maxillary sinus augmentation, the area will be prepared by lifting a full-thickness flap. The sinus membrane will be carefully elevated by opening a window through the lateral wall of the sinus on both sides. Bio-oss bovine bone graft on one side will be placed in the space prepared in the sinus region by random selection. For Platelet-rich fibrin prepared, the blood taken from the patient to a 20 cc injektor was put into titanium tubes and prepared by centrifugation at 2700 rpm for 13 minutes according to the standard protocol. Then, 6 months after the surgery, histological sample will be taken with a trephine bur in both groups and the implant will be placed in accordance with the standard protocol. The stability value (ISQ) of the placed implant will be measured with the Ostell device at the time the implant is placed and 3 months after it is placed.
  Arms: Bio-oss bovine bone graft with maxillary sinus augmentation and implant placement

SUMMARY:
Before placement of the dental implant in the posterior maxilla where the maxillary sinus is pneumatized, it is necessary to elevate of the sinus mucosa from the sinus floor (sinus lift) and to provide new bone formation by using bone-forming graft materials (maxillary sinus augmentation) in the space obtained. In the bilateral maxillary posterior region with insufficient bone height with tooth deficiency, two-stage sinus lift and placement of platelet-rich fibrin prepared with titanium on one side and bovine bone graft on the other side in the implant surgery will affect the primary stability of the implant, the obtained bone histology, volume, height and density is the evaluation of its effect on it. Ten patients who required a maxillary sinus augmentation procedure for implant placement in the bilateral atrophic maxilla were included. Bio-Oss bovine bone graft was made on one side of the patients and randomly assigned to the control group, and the other side was randomly assigned to the test group using platelet-rich fibrin prepared with titanium.

DETAILED DESCRIPTION:
In addition to insufficient bone height with bone resorption of the posterior maxilla after tooth loss, the pneumatization of the maxillary sinus is one of the factors that prevent implant placement in the posterior maxilla. For this, it is necessary to raise the sinus mucosa from the sinus floor (sinus lift) and to provide new bone formation by using bone graft materials (maxillary sinus augmentation) in the resulting sinüs cavity. Two-stage sinus augmentation and implant placement have been recognized as a good clinical model for evaluating the performance of graft materials. Because bone formation takes place in a closed area and with minimal intervention of external factors. Platelet-rich fibrin (T-PRF) prepared with titanium from autologous thrombocyte concentrates showed a tighter polymerized fibrin structure and a long dissolution process, and it was reported that new bone formation started on the 15th day with the placed T-PRF and was effective in 30 days. In a study, comparing the use of allograft and T-PRF in maxillary sinus augmentation, the group in which only T-PRF was applied showed successful clinical and histological results, and new bone formation was accelerated up to 4 months compared to allografts. The primary stability of the implants placed was similar in both groups.

The primary stability of the implant, the bone histology, volume, height and density of the two-stage sinus lift in the bilateral maxillary posterior region with insufficient bone height with tooth deficiency, and the placement of platelet-rich fibrin prepared with titanium on one side and bovine bone graft on the other side in implant surgery, evaluation of its effect.

Bilateral atrophic maxilla dental implant placement and who needed maxillary sinus augmentation, and who did not smoke or smoked at most 10 cigarettes will be included in the study. Before the operation, systemic and dental anamnesis will be taken from the patient and clinical measurements and radiographic images will be recorded.

Inclusion criteria

1. be over 18 years old
2. The patient does not have any systemic disease
3. Patients who do not smoke or smoke less than 10 times a day
4. Patients who need fixed implant supported prosthesis in the bilateral maxillary posterior region
5. Bilateral posterior maxilla residual bone height <5 mm on current radiographs
6. Full mouth plaque insertion and bleeding score ≤15%

Exclusion criteria

1. Being outside the specified age range
2. Patients who smoke more than 10 cigarettes a day
3. History of acute infection or chronic sinusitis in the Schneiderian membrane
4. Having allergies involving the respiratory system
5. Any contraindication for systematic periodontal surgery (Patients with bleeding platelet disorders, bisphosphonate therapy, uncontrolled diabetes (HbA1c > 6%, blood glucose level > 110 mg/dl)),
6. Bilateral posterior maxilla residual bone height >5 mm on current radiographs
7. Full mouth plaque insertion and bleeding score ≥15% Bio-oss bovine bone graft on one side and platelet-rich fibrin prepared with titanium on the other side of 10 patients who require bone height increase with the maxillary sinus augmentation procedure for implant placement in the atrophic posterior maxilla with a bilateral bone height of less than 5 mm will be applied. Test group and Control group will be written in closed envelopes, and platelet-rich fibrin prepared with titanium groups and Bio-oss bovine bone graft will be selected randomly.

The operation date will be given after the patient is given oral hygiene training and 4 weeks after receiving Phase I routine periodontal treatment. The data to be obtained preoperatively and postoperatively are as follows:

1. Plaque index (Löe&Silness): It is obtained by measuring with a periodontal probe from 4 regions of a tooth (mesial, distal, buccal and lingual).
2. Gingival index (Silness&Löe): It is obtained by measuring with a periodontal probe from 4 regions of a tooth (mesial, distal, buccal and lingual).
3. Attachment loss: The distance between the free gingiva and the base of the periodontal sulcus, based on the enamel-cementum boundary of a tooth, is measured using a periodontal probe.
4. Bleeding index on probing (Ainamo & Bay): In this index, probing is performed by gently walking around the pocket. As a result of probing, the evaluation is made by looking at the presence or absence of bleeding in the gingiva. A positive value is given if bleeding occurs within 10-15 seconds after probing in the mesial, distal, buccal and lingual gingival parts of all teeth. The ratio of the bleeding area to the examined area is expressed as %.
5. Pocket depth: It is the vertical distance measured between the base of the periodontal sulcus and the gingival margin with a standard periodontal probe
6. Residual bone height: It is the distance from the top of the alveolar crest to the floor of the maxillary sinus in the preoperative tomography.
7. Sinus mucosal thickness: It is the measurement of the membrane's sinus floor and adjacent surfaces of the sinus cavity. Its thickness varies between 2.16-3.11.
8. Sinus volume: It is the measurement of the vertical and horizontal heights of the sinus cavity.
9. Fractal analysis: By placing circles of various diameters randomly in the image, the pixels of the image border inside the circles are counted. It is stated that it reflects changes in trabecular bone density and mineral loss in bone. When the panoramic radiographs were examined with fractal analysis, it was stated that the increase in the fractal size of the bone around the implant correlated with successful osteointegration and healing of the trabecular bone.
10. Hounsfield unit: System computers assign a number to all voxels in the images obtained by computed tomography according to this scale. It is to paint voxels that have received numerical values with black, white and gray tones in between that match the numbers they receive. Changes in bone can be observed

ELIGIBILITY:
Inclusion Criteria:

1. >18 years old
2. The patient does not have any systemic disease
3. Patients who need fixed implant-supported prosthesis in the bilateral maxillary posterior region
4. Bilateral posterior maxilla residual bone height <5 mm
5. Full mouth plaque and bleeding score ≤15%

Exclusion Criteria:

1. Patients who smoke more than 10 cigarettes a day
2. History of acute infection or chronic sinusitis in the Schneiderian membrane
3. Having allergies involving the respiratory system
4. Any contraindication for systematic periodontal surgery (Patients with bleeding platelet disorders, bisphosphonate therapy, uncontrolled diabetes (HbA1c > 6%, blood glucose level > 110 mg/dl)),
5. Bilateral posterior maxilla residual bone height >5 mm

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-03-14 (Actual); Primary Completion 2023-04-14 (Actual); Study Completion 2023-04-14 (Actual)

PRIMARY OUTCOMES:
Bone gain change radiologically | Postoperatively 6th month
  Change of the distance from the top of the alveolar crest to the floor of the maxillary sinus in the cone beam computerized tomography at between baseline and postoperatively 6th month.
Histomorphometric bone changes | Postoperatively 6th month
  Following at 6th month from sinus augmentation, histological samples will be evaluated new bone formation.

SECONDARY OUTCOMES:
Bone density changes | Postoperatively 6th month
  Bone density will be evaluated on cone beam computerized tomography at 6 months after surgery with Hounsfield Units.
  Primary stability 3 months after implant placement (T2): Resonance frequency analysis is the unit of measurement in determining the stability of the implant. It gives the resonance frequency (kHz) on a clinically usable scale from 1-100 ISQ. It will be measured 3 months after the implant is placed.
  Sinus volume change (T0-T1): The measurement of the vertical and horizontal heights of the sinus cavity on tomography before and 6 months after surgery will be compared.
Primary Stabilization Value | Immediately after dental implant placement,
  Resonance frequency analysis is the unit of measurement in determining the stability of the implant. It gives the resonance frequency (kHz) on a clinically usable scale from 1-100 ISQ.
Secondary Implant Stabilization | At healing cap session, following dental implant placement 3rd month
  Resonance frequency analysis is the unit of measurement in determining the stability of the implant. It gives the resonance frequency (kHz) on a clinically usable scale from 1-100 ISQ.

CONTACTS AND LOCATIONS:
Overall Officials: Berceste Güler, Study Director — Kütahya Health Sciences University
Locations (1):
- Kütahya Health Sciences University Faculty of Dentistry, Department of Periodontology, Kütahya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data can be shared if the principal investigator is contacted
Supporting Information: CSR
Time Frame: Following acceptance of manuscript
Access Criteria: Individual participant data can be shared if the principal investigator is contacted

REFERENCES:
- [Result] Irinakis T. Efficacy of injectable demineralized bone matrix as graft material during sinus elevation surgery with simultaneous implant placement in the posterior maxilla: clinical evaluation of 49 sinuses. J Oral Maxillofac Surg. 2011 Jan;69(1):134-41. doi: 10.1016/j.joms.2010.07.028. Epub 2010 Nov 2. PMID 21050634
- [Result] Corbella S, Taschieri S, Del Fabbro M. Long-term outcomes for the treatment of atrophic posterior maxilla: a systematic review of literature. Clin Implant Dent Relat Res. 2015 Feb;17(1):120-32. doi: 10.1111/cid.12077. Epub 2013 May 8. PMID 23656352
- [Result] Adali E, Yuce MO, Gunbay T, Gunbay S. Does Concentrated Growth Factor Used With Allografts in Maxillary Sinus Lifting Have Adjunctive Benefits? J Oral Maxillofac Surg. 2021 Jan;79(1):98-108. doi: 10.1016/j.joms.2020.07.217. Epub 2020 Aug 5. PMID 32866488
- [Result] Tunali M, Ozdemir H, Kucukodaci Z, Akman S, Yaprak E, Toker H, Firatli E. A novel platelet concentrate: titanium-prepared platelet-rich fibrin. Biomed Res Int. 2014;2014:209548. doi: 10.1155/2014/209548. Epub 2014 Jan 21. PMID 24563860
- [Result] Olgun E, Ozkan SY, Atmaca HT, Yalim M, Hendek MK. Comparison of the clinical, radiographic, and histological effects of titanium-prepared platelet rich fibrin to allograft materials in sinus-lifting procedures. J Investig Clin Dent. 2018 Nov;9(4):e12347. doi: 10.1111/jicd.12347. Epub 2018 Jun 12. PMID 29893477
- [Derived] Eken S, Guler Ayyildiz B, Altay B, Ari NS, Ozatik O. Clinical, Radiological, and Histomorphometric Comparison of the Use of Deproteinized Bovine Bone Mineral and Titanium-Prepared Platelet-Rich Fibrin in Maxillary Sinus Augmentation: A Split-Mouth Randomized Controlled Clinical Study. J Oral Maxillofac Surg. 2025 Mar;83(3):322-331. doi: 10.1016/j.joms.2024.11.006. Epub 2024 Nov 19. PMID 39638292